CLINICAL TRIAL: NCT05903183
Title: A Phase 2a Randomized, Observer-blind, Placebo-controlled, Dosage Optimization, Multi-center Clinical Trial to Evaluate the Safety and Immunogenicity of IVX-A12, a Respiratory Syncytial Virus and Human Metapneumovirus Bivalent Combination Virus-like Particle Protein Subunit Vaccine, in Adults 60 to 85 Years of Age
Brief Title: A Study to Evaluate the Safety and Immunogenicity of IVX-A12 in Participants of 60 to 85 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icosavax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ICVX-12-201
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Respiratory syncytial virus (RSV); Human metapneumovirus (hMPV); Bivalent virus-like particle protein subunit vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IVX-A12 Vaccine Formulation 1 (Experimental): Participants will receive a single dose of IVX-A12 intramuscular (IM) injection on Day 0.
  Interventions: Biological: IVX-A12
- IVX-A12 Vaccine Formulation 2 (Experimental): Participants will receive a single dose of IVX-A12 IM injection on Day 0.
  Interventions: Biological: IVX-A12
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo IM injection on Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IVX-A12 — IVX-A12 without adjuvant
  Arms: IVX-A12 Vaccine Formulation 1
Biological: IVX-A12 — IVX-A12 with adjuvant
  Arms: IVX-A12 Vaccine Formulation 2
Biological: Placebo — Diluent
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to assess the safety, tolerability and immunogenicity of a bivalent respiratory syncytial virus (RSV)/human metapneumovirus (hMPV) virus-like particle (VLP) candidate vaccine (IVX-A12) compared to placebo, when administered as a single-dose regimen in healthy older adults 60 to 85 years of age.

DETAILED DESCRIPTION:
The IVX-A12 Phase 2a clinical trial is a randomized, observer-blind, placebo-controlled, dosage optimization, multi-center trial to evaluate the safety and immunogenicity of a single intramuscular (IM) dose of IVX-A12, with or without adjuvant, in adults 60 to 85 years of age.

Participants will be administered a single shot of IVX-A12, at specified dosage levels, or placebo. The overall duration of the study is up to 1 year (12 months). A subset of participants will be followed for an additional 12 months for a total duration of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, who must be in stable health based on medical history, vital signs, physical examination, and laboratory evaluation prior to vaccination, in the investigator's clinical judgment
2. Participants may have ongoing chronic conditions (comorbidities such as hypertension, congestive heart failure, chronic obstructive pulmonary disease, type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism) who are, in the investigator's opinion, medically compensated and without recent exacerbation within the prior 3 months
3. Participants able to voluntarily give written informed consent and can comply with trial procedures including follow-up for approximately 12 months after vaccination
4. Body mass index 17 to less than (<) 40 kilograms per square meter (kg/m^2) at screening
5. Before randomization, female participants must be unable to conceive (example, menopausal, that is, 12 consecutive months without menstruation, hysterectomy, oophorectomy, etc.) and not intending to conceive by any method
6. Participants must agree not to donate blood from the time of vaccination through 3 months after vaccination
7. Participants must be willing to provide verifiable identification and have the means to be contacted and to contact the investigator or the site's staff during the entire clinical trial

Exclusion Criteria:

1. Participants with moderate or severe liver disease, metastatic solid tumor, and acquired immunodeficiency syndrome (AIDS) are to be excluded. In addition, participants with underlying significant illness or condition(s) or ongoing treatment that, in the opinion of the investigator, could (i) interfere with the conduct of the trial, (ii) pose an unacceptable risk to the participant in this trial, (iii) interfere with the participant's ability to comply with the trial procedures or abide by the procedures
2. Older adults who meet frail elderly criteria (older persons with medical, nutritional, cognitive, emotional, or activity impairments, as defined by the Dalhousie Clinical Frailty Score greater than or equal to [>=]4)
3. Prior receipt of any licensed or investigational RSV or hMPV vaccine within the past 12 months
4. Prior receipt of another investigational medicinal product (IMP; trial drug, biologic, or device) not authorized for use in the United States of America (USA) and European Union within the past 3 months
5. Laboratory-confirmed RSV or hMPV infection within 12 months prior to enrollment
6. Currently enrolled or plan to participate in another clinical trial with an investigational agent (including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) to be received during the trial period
7. History of malignancy within 5 years before screening not in the following categories: (i) participants with squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix may be enrolled at the discretion of the investigator, (ii) participants with a history of malignancy within 5 years before screening, with minimal risk of recurrence per investigator's judgment, can be enrolled
8. Acute illness, with or without fever at the time of planned vaccination
9. History of hypersensitivity or serious adverse reactions to vaccines, such as anaphylaxis or angioedema, or any known allergies to any component of the IVX-121 and/or IVX-241 vaccine, or hypersensitivity to latex
10. Abnormal function of the immune system resulting from clinical conditions including chronic administration of systemic corticosteroids (oral/intravenous/IM at a daily dose equivalent of greater than (>) 20 milligram (mg) prednisone in a period of more than 14 days), or administration of immunosuppressive chemotherapy, biologics, or radiotherapy within the past 3 months prior to planned vaccination
11. Participants who have received treatment with immunoglobulins or other biologics, such as immunosuppressive therapies expected to modify immune response to vaccination (including monoclonal antibodies [MAbs] for chronic underlying conditions) within the past 3 months prior to planned vaccination
12. Trial personnel as an immediate family or household member
13. For licensed vaccines:

    1. Receipt of licensed inactivated vaccines (including seasonal influenza vaccine) within 14 days prior to trial vaccine administration on Day 0, or licensed replicating vaccines such as ribonucleic acid (RNA) or live-attenuated virus vaccines within 30 days prior to Day 0
    2. Receipt of licensed vaccines is permitted after completion of the Day 28 visit
    3. Receipt of any licensed Coronavirus Disease-2019 (COVID-19) vaccines is permitted if dosing regimen completed within 21 days prior to Day 0 or after completion of the Day 28 visit.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - AMR Phoenix, Tempe, Arizona
  - Cenexel RCA, Hollywood, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Velocity Clinical Research-Boise, Meridian, Idaho
  - ASR, LLC, Nampa, Idaho
  - Johnson City Clin-Trials (JCCT), Lenexa, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Velocity Clinical Research, Omaha, Nebraska
  - Rochester Clinical Research, Inc, Rochester, New York
  - PanAmerican Clinical Research, Brownsville, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ICVX-12-201&attachmentIdentifier=87148cb9-99d7-49de-b512-993369bc114d&fileName=ICVX-12-201_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ICVX-12-201&attachmentIdentifier=ecedb9ce-bd92-4ffe-ac0d-00f7c1a7e9d5&fileName=ICVX-12-201_Redacted_SAP.pdf&versionIdentifier=
- See also: ICVX-12-201_Redacted CSR_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ICVX-12-201&attachmentIdentifier=eb2ddeaa-ee6e-4b60-88a4-dc27f97b896a&fileName=ICVX-12-201_Redacted_CSR_synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 10 investigative sites in the United States.
Pre-assignment Details: A total 264 participants were enrolled and randomized to receive vaccinations in this study. The study has a Main Trial part and Observation Extension Trial part.
Groups:
- Main Trial Part: IVX-A12 150 mcg: Participants received a single dose of 150 mcg IVX-A12, IM injection on Day 1.
- Main Trial Part: IVX-A12 150 mcg With MF59: Participants received a single dose of 150 mcg IVX-A12 adjuvanted with MF59, IM injection on Day 1.
- Main Trial Part: Placebo: Participants received matching placebo on Day 1.
- Observational Extension Part: IVX-A12 150 mcg: Participants who received a single dose of 150 mcg IVX-A12, IM injection on Day 1 in Main Trial part were enrolled and observed in Extension part.
- Observational Extension Part: Placebo: Participants who received matching placebo on Day 1 in Main Trial part were enrolled and observed in Extension part.
Period: Main Trial Part (365 Days)
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo | Observational Extension Part: IVX-A12 150 mcg | Observational Extension Part: Placebo
Started | 102 | 109 | 53 | 0 | 0
Safety Set | 103 (One participant was randomized in IVX-A12 150 mcg with MF59 group but was treated in IVX-A12 150 mcg group.) | 108 (One participant was randomized in IVX-A12 150 mcg with MF59 group but was treated in IVX-A12 150 mcg group.) | 53 | 0 | 0
Completed | 99 | 107 | 51 | 0 | 0
Not Completed | 3 | 2 | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Observation Extension Part (144 Days)
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo | Observational Extension Part: IVX-A12 150 mcg | Observational Extension Part: Placebo
Started | 0 | 0 | 0 | 35 (Participants who completed the main part and gave consent to enroll in the extension part were included.) | 20 (Participants who completed the main part and gave consent to enroll in the extension part were included.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 35 | 20
Not completed — Sponsor's decision | 0 | 0 | 0 | 35 | 20

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all randomized participants who received a dose of IVX-A12 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo | Total
Number analyzed (Participants) | 102 | 109 | 53 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (6.05) | 69.3 (5.83) | 68.8 (5.79) | 69.2 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 65 | 32 | 152
  Male | 47 | 44 | 21 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 7 | 49
  Not Hispanic or Latino | 82 | 84 | 46 | 212
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 12 | 14 | 5 | 31
  White | 88 | 94 | 48 | 230
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Reactions (ARs) and Systemic ARs
Description: Solicited local ARs include pain, tenderness, erythema, and swelling. Solicited systemic ARs include headache, chills, fatigue, myalgia, arthralgia, vomiting, diarrhea, and fever.
Time Frame: From Day 0 to Day 6
Population: The Safety Set includes all participants who received any amount of IVX-A12 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 103 | 108 | 53
Participants
  Solicited Local Adverse Reactions | 46 | 68 | 5
  Solicited Systemic Adverse Reactions | 34 | 56 | 19

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An unsolicited AE is an AE that was not solicited using the post-vaccination diary and that was spontaneously communicated by a participant.
Time Frame: From Day 0 to Day 28
Population: The Safety Set includes all participants who received any amount of IVX-A12 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 103 | 108 | 53
Participants | 33 | 38 | 13

3. Primary Outcome: Model-adjusted Geometric Mean Titers (GMT) for RSV-A, RSV-B, hMPV-A, and hMPV-B-specific Neutralizing Antibodies (NAb)
Description: Model-adjusted GMT and corresponding 95% CI were derived from an analysis of covariance (ANCOVA) model of log2 titer at Day 28 with independent variables of log2 baseline titer, age group, and treatment group.
Time Frame: At Day 28
Population: The PPS includes all participants in the FAS who received a dose of IVX-A12 or placebo and have no major protocol deviations, which may exclude participants from PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: MN50 titer
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
MN50 titer
  RSV-A | 11980.96 [9760.34 to 14706.80] | 11167.48 [9101.24 to 13702.82] | 1944.00 [1449.07 to 2607.97]
  RSV-B | 7787.22 [6516.69 to 9305.46] | 6560.64 [5493.69 to 7834.81] | 2205.65 [1708.45 to 2847.55]
  hMPV-A | 1643.58 [1378.03 to 1960.31] | 1416.79 [1187.96 to 1689.69] | 465.09 [361.26 to 598.76]
  hMPV-B | 15503.09 [13515.07 to 17783.54] | 17317.65 [15103.86 to 19855.92] | 6370.00 [5230.31 to 7758.03]

4. Primary Outcome: Model-adjusted Geometric Mean Concentrations (GMC) for RSV and hMPV Prefusion F Protein-specific IgG Antibodies (Ab)
Description: Model-adjusted GMC and corresponding 95% CI were derived from an analysis of covariance (ANCOVA) model of log2 concentration at Day 28 with independent variables of log2 baseline concentration, age group, and treatment group.
Time Frame: At Day 28
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter (EU/mL)
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
ELISA units per milliliter (EU/mL)
  RSV | 1549.06 [1369.32 to 1752.38] | 1556.06 [1375.49 to 1760.33] | 393.03 [329.37 to 468.99]
  hMPV | 1707.15 [1482.99 to 1965.19] | 1856.88 [1614.14 to 2136.12] | 444.74 [363.06 to 544.79]

5. Primary Outcome: Percentage of Participants With a >=4-fold Increase in Serum RSV-A, RSV-B, hMPV-A, and hMPV-B-specific NAb Titers
Description: Proportion of participants with non-missing results at the specified visit achieving a 4-fold or greater increase in NAb titer versus baseline (Day 0).
Time Frame: From Day 0 (pre-vaccination) up to Day 28 post-vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
percentage of participants
  RSV-A: Day 28 | 57.3 | 55.1 | 0
  RSV-B: Day 28 | 43.8 | 36.7 | 2.1
  hMPV-A: Day 28 | 38.5 | 28.6 | 0.0
  hMPV-B: Day 28 | 25.0 | 35.7 | 0

6. Primary Outcome: Percentage of Participants With >=4-fold Increase in RSV and hMPV-specific IgG Ab Concentration
Description: Proportion of participants with non-missing results at the specified visit achieving a 4-fold or greater increase in Ab concentration versus baseline (Day 0).
Time Frame: From Day 0 (pre-vaccination) up to Day 28 post-vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
percentage of participants
  RSV: Day 28 | 45.8 | 42.9 | 0.0
  hMPV: Day 28 | 47.9 | 52.0 | 0.0

7. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Serum for RSV-A, RSV-B, hMPV-A, and hMPV-B-Specific NAb Titers
Description: GMFR is defined as the geometric mean of the ratio of NAb titer at specified timepoints after vaccination divided by baseline (Day 0) titer.
Time Frame: From Day 0 (pre-vaccination) up to Day 28 post-vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
fold rise
  RSV-A: Day 28 | 5.86 [4.59 to 7.48] | 5.07 [3.92 to 6.57] | 0.95 [0.85 to 1.06]
  RSV-B: Day 28 | 3.67 [2.99 to 4.50] | 3.11 [2.54 to 3.80] | 1.08 [0.87 to 1.34]
  hMPV-A: Day 28 | 3.150 [2.544 to 3.900] | 2.486 [2.022 to 3.058] | 0.910 [0.764 to 1.083]
  hMPV-B: Day 28 | 2.426 [2.016 to 2.919] | 2.746 [2.254 to 3.346] | 0.936 [0.806 to 1.087]

8. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Serum for RSV and hMPV Prefusion F Protein-specific IgG Ab Concentrations
Description: GMFR is defined as the geometric mean of the ratio of Ab concentration at specified timepoints after vaccination divided by baseline (Day 0) concentration.
Time Frame: From Day 0 (pre-vaccination) up to Day 28 post-vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
fold rise
  RSV: Day 28 | 3.858 [3.253 to 4.575] | 3.465 [2.896 to 4.146] | 0.987 [0.917 to 1.063]
  hMPV: Day 28 | 4.008 [3.321 to 4.838] | 4.266 [3.561 to 5.111] | 0.896 [0.775 to 1.037]

9. Secondary Outcome: Number of Participants With Serious Adverse Event (SAE), Medically-attended Adverse Events (MAAEs), and AEs Leading to Trial Withdrawal
Description: An SAE is defined as any untoward medical occurrence that met one or more of the following: resulted in death; was immediately life-threatening; required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly or birth defect in the offspring of a subject; was an important and significant medical event that might have jeopardized the participant or required medical intervention to prevent one of the aforementioned outcomes. Any AESI occurring during the trial will be categorized and reported as an SAE. These AESIs include anaphylaxis, thrombocytopenia, and other potential immune-mediate conditions (including Guillain Barre syndrome). MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From Day 0 up to the end of study (up to Day 365)
Population: The Safety Set includes all participants who received any amount of IVX-A12 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 103 | 108 | 53
Participants
  SAEs | 5 | 3 | 1
  MAAEs | 54 | 60 | 21
  AE Leading to Study Discontinuation | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe Lower Respiratory Tract Illness (LRTI) Caused by RSV and/or hMPV
Description: Data is summarized as the number of subjects with at least one LRTI event (mild, moderate, or severe) by treatment group.
Time Frame: From Day 0 up to Day 365 (end of study)
Population: The Safety Set includes all participants who received any amount of IVX-A12 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 103 | 108 | 53
Participants | 4 | 2 | 0

11. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe LRTI Cases Not Caused by RSV or hMPV
Description: as for outcome 10
Time Frame: From Day 0 up to Day 365 (end of study)
Population: The Safety Set includes all participants who received any amount of IVX-A12 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 103 | 108 | 53
Participants | 14 | 11 | 4

12. Secondary Outcome: Number of Participants With Clinically Significant Safety Laboratory Parameters
Time Frame: At Screening, Days 0, 7 and 28
Population: The Safety Set includes all participants who received any amount of IVX-A12 or placebo.
Measure: Number; unit: participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 103 | 108 | 53
participants | 0 | 0 | 0

13. Secondary Outcome: Model-Adjusted GMTs for RSV-A, RSV-B, hMPV-A, and hMPV-B-specific NAb
Description: Model-adjusted GMT and corresponding 95% CI were derived from an analysis of covariance (ANCOVA) model of log2 titer at each post-baseline timepoint with independent variables of log2 baseline titer, age group, and treatment group.
Time Frame: At Days 180 and 365
Population: The PPS includes all participants in the FAS who received a dose of IVX-A12 or placebo and have no major protocol deviations, which may exclude participants from PPS. Here 'n' refers to number of participants analyzed at given timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: MN50 titer
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
MN50 titer
  RSV-A: Day 180: number analyzed (Participants) | 92 | 92 | 45
  RSV-A: Day 180 | 6864.00 [5643.98 to 8347.73] | 7145.43 [5857.89 to 8715.98] | 2741.63 [2068.75 to 3633.36]
  RSV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-A: Day 365 | 4142.06 [3464.80 to 4951.71] | 3793.79 [3164.62 to 4548.04] | 1933.12 [1500.23 to 2490.90]
  RSV-B: Day 180: number analyzed (Participants) | 93 | 91 | 45
  RSV-B: Day 180 | 4536.59 [3856.59 to 5336.50] | 4152.76 [3516.39 to 4904.29] | 2205.81 [1744.68 to 2788.83]
  RSV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-B: Day 365 | 2690.13 [2306.79 to 3137.18] | 2640.17 [2124.78 to 3085.15] | 1640.56 [1318.92 to 2040.65]
  hMPV-A: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-A: Day 180 | 667.67 [582.87 to 764.80] | 690.94 [601.39 to 793.83] | 383.31 [315.11 to 466.27]
  hMPV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-A: Day 365 | 589.68 [508.98 to 683.17] | 535.25 [460.94 to 621.53] | 421.28 [341.91 to 519.08]
  hMPV-B: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-B: Day 180 | 9709.73 [8393.50 to 11232.35] | 9482.90 [8175.75 to 10999.05] | 4243.59 [3437.19 to 5239.18]
  hMPV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-B: Day 365 | 8519.18 [7290.09 to 9955.49] | 7699.03 [6574.90 to 9015.36] | 4743.25 [3800.77 to 5919.44]

14. Secondary Outcome: Model-Adjusted GMCs for RSV and hMPV Prefusion F Protein-specific IgG Ab Concentrations
Description: Model-adjusted GMC and corresponding 95% CI were derived from an analysis of covariance (ANCOVA) model of log2 concentration at each post-baseline timepoint with independent variables of log2 baseline concentration, age group, and treatment group.
Time Frame: At Days 180, and 365
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter (EU/mL)
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
ELISA units per milliliter (EU/mL)
  RSV: Day 180: number analyzed (Participants) | 93 | 92 | 45
  RSV: Day 180 | 730.14 [640.20 to 832.72] | 739.32 [646.32 to 845.70] | 313.74 [259.41 to 379.45]
  RSV: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV: Day 365 | 781.54 [704.30 to 867.24] | 772.83 [695.20 to 859.12] | 406.42 [350.62 to 471.11]
  hMPV: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV: Day 180 | 925.81 [811.73 to 1055.92] | 937.01 [819.77 to 1071.02] | 386.81 [319.62 to 468.12]
  hMPV: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV: Day 365 | 1018.26 [909.04 to 1140.59] | 994.03 [886.24 to 1114.94] | 560.77 [476.93 to 659.35]

15. Secondary Outcome: Percentage of Participants With a >=4-fold Increase in Serum RSV-A, RSV-B, hMPV-A, and hMPV-B-specific NAb Titers
Description: as for outcome 5
Time Frame: From Day 0 (pre-vaccination) up to Day 180 and Day 365 post-vaccination
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
percentage of participants
  RSV-A: Day 180: number analyzed (Participants) | 92 | 92 | 45
  RSV-A: Day 180 | 35.9 | 35.9 | 6.7
  RSV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-A: Day 365 | 18.2 | 21.6 | 2.3
  RSV-B: Day 180: number analyzed (Participants) | 93 | 91 | 45
  RSV-B: Day 180 | 23.7 | 18.7 | 4.4
  RSV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-B: Day 365 | 6.8 | 9.1 | 2.3
  hMPV-A: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-A: Day 180 | 7.5 | 6.5 | 0.0
  hMPV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-A: Day 365 | 6.8 | 4.5 | 2.3
  hMPV-B: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-B: Day 180 | 12.9 | 14.1 | 0.0
  hMPV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-B: Day 365 | 9.1 | 3.4 | 0.0

16. Secondary Outcome: Percentage of Participants With >=4-fold Increase in RSV and hMPV Prefusion F Protein-specific IgG Ab Concentrations
Description: as for outcome 6
Time Frame: From Day 0 (pre-vaccination) up to Days 180, and 365 post-vaccination
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
percentage of participants
  RSV: Day 180: number analyzed (Participants) | 93 | 92 | 45
  RSV: Day 180 | 12.9 | 12.0 | 0.0
  RSV: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV: Day 365 | 8.0 | 10.2 | 0.0
  hMPV: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV: Day 180 | 21.5 | 19.6 | 0.0
  hMPV: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV: Day 365 | 27.3 | 20.5 | 0.0

17. Secondary Outcome: Percentage of Participants With a >=8-fold Increase in Serum RSV-A, RSV-B, hMPV-A, and hMPV-B-specific NAb Titers
Description: Proportion of participants with non-missing results at the specified visit achieving a 8-fold or greater increase in NAb titer versus baseline (Day 0).
Time Frame: From Day 0 (pre-vaccination) up to Days 28, 180, and 365 post-vaccination
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
percentage of participants
  RSV-A: Day 28 | 39.6 | 38.8 | 0.0
  RSV-A: Day 180: number analyzed (Participants) | 92 | 92 | 45
  RSV-A: Day 180 | 16.3 | 20.7 | 2.2
  RSV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-A: Day 365 | 8.0 | 9.1 | 0.0
  RSV-B: Day 28 | 21.9 | 16.3 | 2.1
  RSV-B: Day 180: number analyzed (Participants) | 93 | 91 | 45
  RSV-B: Day 180 | 7.5 | 4.4 | 0.0
  RSV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-B: Day 365 | 2.3 | 3.4 | 0.0
  hMPV-A: Day 28 | 13.5 | 15.3 | 0
  hMPV-A: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-A: Day 180 | 2.2 | 2.2 | 0
  hMPV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-A: Day 365 | 1.1 | 0 | 0
  hMPV-B: Day 28 | 11.5 | 19.4 | 0
  hMPV-B: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-B: Day 180 | 4.3 | 4.3 | 0
  hMPV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-B: Day 365 | 1.1 | 2.3 | 0

18. Secondary Outcome: GMFR in Serum for RSV-A, RSV-B, hMPV-A, and hMPV-B-specific NAb Titers and RSV and hMPV Prefusion F Protein-specific IgG Ab Concentrations
Description: as for outcome 8
Time Frame: From Day 0 (pre-vaccination) up to Day 180 and Day 365 post-vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
fold rise
  RSV-A: Day 180: number analyzed (Participants) | 92 | 92 | 45
  RSV-A: Day 180 | 3.21 [2.66 to 3.88] | 3.18 [2.44 to 4.15] | 1.34 [1.09 to 1.65]
  RSV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-A: Day 365 | 1.97 [1.63 to 2.39] | 1.68 [1.33 to 2.13] | 0.94 [0.78 to 1.13]
  RSV-B: Day 180: number analyzed (Participants) | 93 | 91 | 45
  RSV-B: Day 180 | 2.02 [1.67 to 2.45] | 1.88 [1.55 to 2.29] | 1.02 [0.80 to 1.29]
  RSV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-B: Day 365 | 1.23 [1.02 to 1.47] | 1.20 [0.99 to 1.45] | 0.76 [0.61 to 0.94]
  hMPV-A: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-A: Day 180 | 1.285 [1.079 to 1.530] | 1.115 [0.909 to 1.367] | 0.736 [0.562 to 0.962]
  hMPV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-A: Day 365 | 1.094 [0.914 to 1.310] | 0.866 [0.706 to 1.063] | 0.793 [0.606 to 1.037]
  hMPV-B: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-B: Day 180 | 1.482 [1.258 to 1.747] | 1.456 [1.210 to 1.753] | 0.622 [0.500 to 0.773]
  hMPV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-B: Day 365 | 1.262 [1.056 to 1.509] | 1.153 [0.961 to 1.384] | 0.681 [0.551 to 0.841]
  RSV Pre-F: Day 180: number analyzed (Participants) | 93 | 92 | 45
  RSV Pre-F: Day 180 | 1.728 [1.487 to 2.007] | 1.638 [1.380 to 1.945] | 0.774 [0.665 to 0.901]
  RSV Pre-F: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV Pre-F: Day 365 | 1.844 [1.631 to 2.084] | 1.687 [1.457 to 1.952] | 0.973 [0.874 to 1.084]
  hMPV Pre-F: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV Pre-F: Day 180 | 2.157 [1.822 to 2.553] | 2.118 [1.786 to 2.512] | 0.794 [0.691 to 0.912]
  hMPV Pre-F: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV Pre-F: Day 365 | 2.380 [2.029 to 2.792] | 2.293 [1.989 to 2.644] | 1.149 [0.986 to 1.339]

19. Secondary Outcome: Reverse Cumulative Distribution (RCD) Curve of Serum NAb Titers and IgG Ab Concentrations
Description: The median, as well as 25th and 75th percentiles of serum NAb titers and IgG Ab concentrations are summarized at specified timepoints.
Time Frame: At Days 28, 180, and 365 post-vaccination
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: MN50 titer
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo
Number analyzed (Participants) | 96 | 98 | 47
MN50 titer
  RSV-A: Day 0 | 1779.18 [894.07 to 3661.52] | 2068.22 [984.30 to 4601.80] | 1764.10 [765.60 to 4136.50]
  RSV-A: Day 28 | 12010.69 [4870.35 to 23207.12] | 10806.21 [4939.50 to 25893.80] | 1943.00 [772.80 to 3576.80]
  RSV-A: Day 180: number analyzed (Participants) | 92 | 92 | 45
  RSV-A: Day 180 | 6393.44 [3098.72 to 11645.52] | 6244.78 [3200.74 to 14601.61] | 2601.00 [861.10 to 5542.70]
  RSV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-A: Day 365 | 3793.15 [1869.68 to 6393.49] | 3630.01 [1828.40 to 8923.32] | 1769.58 [852.51 to 3427.73]
  RSV-B: Day 0 | 1965.30 [974.83 to 4937.85] | 2046.80 [1068.30 to 4611.8] | 1722.20 [814.40 to 4421.90]
  RSV-B: Day 28 | 6945.86 [3691.86 to 17581.86] | 6491.77 [2957.70 to 13097.10] | 1757.20 [888.60 to 4941.80]
  RSV-B: Day 180: number analyzed (Participants) | 93 | 91 | 45
  RSV-B: Day 180 | 4226.30 [2123.40 to 10341.40] | 3427.10 [1924.60 to 7152.40] | 2192.40 [971.10 to 4308.00]
  RSV-B: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV-B: Day 365 | 2606.69 [1451.24 to 5158.12] | 2191.31 [1365.43 to 5447.75] | 1416.93 [641.92 to 2867.91]
  hMPV-A: Day 0 | 415.73 [264.05 to 816.11] | 538.90 [313.30 to 1068.70] | 360.50 [221.40 to 842.00]
  hMPV-A: Day 28 | 3.145 [1.479 to 5.837] | 2.223 [1.303 to 4.294] | 0.999 [0.643 to 1.306]
  hMPV-A: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV-A: Day 180 | 636.90 [360.30 to 995.40] | 716.65 [450.90 to 1159.94] | 320.50 [220.70 to 677.80]
  hMPV-A: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV-A: Day 365 | 518.85 [312.16 to 810.61] | 514.09 [299.03 to 919.90] | 313.65 [225.71 to 736.60]
  RSV Pre F: Day 0 | 359.94 [222.96 to 694.54] | 432.69 [257.70 to 802.60] | 489.60 [184.50 to 662.60]
  RSV Pre F: Day 28 | 1544.51 [1008.49 to 2328.19] | 1574.69 [1095.80 to 2313.40] | 439.00 [191.80 to 675.90]
  RSV Pre F: Day 180: number analyzed (Participants) | 93 | 92 | 45
  RSV Pre F: Day 180 | 653.30 [437.50 to 1142.20] | 774.70 [499.56 to 1176.65] | 308.60 [133.00 to 628.50]
  RSV Pre F: Day 365: number analyzed (Participants) | 88 | 88 | 44
  RSV Pre F: Day 365 | 691.49 [499.49 to 1105.17] | 879.79 [521.74 to 1355.85] | 483.45 [210.38 to 730.11]
  hMPV Pre F: Day 0 | 410.74 [226.27 to 726.27] | 524.42 [246.20 to 757.90] | 531.20 [273.20 to 855.40]
  hMPV Pre F: Day 28 | 1857.88 [986.18 to 2815.41] | 1757.83 [1275.90 to 2744.10] | 444.00 [254.40 to 851.90]
  hMPV Pre F: Day 180: number analyzed (Participants) | 93 | 92 | 45
  hMPV Pre F: Day 180 | 959.30 [585.40 to 1548.40] | 920.64 [520.62 to 1585.77] | 383.20 [251.40 to 672.30]
  hMPV Pre F: Day 365: number analyzed (Participants) | 88 | 88 | 44
  hMPV Pre F: Day 365 | 967.80 [664.70 to 1543.22] | 989.21 [684.24 to 1632.10] | 621.84 [363.65 to 950.72]

ADVERSE EVENTS:
Time Frame: From study start to end of observational extension part (up to Day 509)
Arm/Group | Main Trial Part: IVX-A12 150 mcg | Main Trial Part: IVX-A12 150 mcg With MF59 | Main Trial Part: Placebo | Observational Extension Part: IVX-A12 150 mcg | Observational Extension Part: Placebo
All-Cause Mortality (participants affected / at risk) | 1/103 | 0/108 | 0/53 | 0/35 | 0/20
Serious Adverse Events (participants affected / at risk) | 5/103 | 3/108 | 1/53 | 1/35 | 0/20
Other Adverse Events (participants affected / at risk) | 75/103 | 81/108 | 42/53 | 3/35 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Trial Part: IVX-A12 150 mcg (N=103) | Main Trial Part: IVX-A12 150 mcg With MF59 (N=108) | Main Trial Part: Placebo (N=53) | Observational Extension Part: IVX-A12 150 mcg (N=35) | Observational Extension Part: Placebo (N=20)
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Stag horn calculus (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Trial Part: IVX-A12 150 mcg (N=103) | Main Trial Part: IVX-A12 150 mcg With MF59 (N=108) | Main Trial Part: Placebo (N=53) | Observational Extension Part: IVX-A12 150 mcg (N=35) | Observational Extension Part: Placebo (N=20)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 6 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 18 | 7 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 6 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 6 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 17 | 8 | 0 | 0
Rhinovirus infection (Infections and infestations) | 9 | 8 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 11 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 9 | 8 | 0 | 0
Fatigue (General disorders) | 8 | 13 | 7 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 6 | 0 | 0 | 0
Blood pressure increased (Investigations) | 2 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 5 | 2 | 0 | 0
Hypertension (Vascular disorders) | 8 | 9 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 13 | 15 | 9 | 0 | 0
Respiratory tract infection (Infections and infestations) | 7 | 12 | 5 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 2 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 3 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 3 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 5 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
HCoV-OC43 infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal cobble stone mucosa (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
HCoV-229E infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 0 | 0
Influenza like illness (General disorders) | 1 | 3 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Effusion (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tardive dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 3 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Device physical property issue (Product Issues) | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Stag horn calculus (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tooth erosion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Human metapneumovirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Renal function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 4 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT05903183/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT05903183/SAP_001.pdf